CLINICAL TRIAL: NCT07072780
Title: Effectiveness of a Novel Low-level Laser Therapy Protocol in Managing Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jin A Yoon, MD, Ph.D, Associate Professor, Department of Rehabilitation Medicine, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-2310-029-132
Record Dates: First submitted 2025-06-20; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Low-level laser therapy; LLLT; Photobiomodulation; Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 904nm LLLT (LTU-904) (Experimental): Participants will receive low-level laser therapy using the LTU-904 device at a wavelength of 904 nm after complex decongestive physiotherapy (CDPT), which includes manual lymphatic drainage, remedial exercises, and intermittent pneumatic compression.
  Interventions: Device: Low-Level Laser Therapy (650 nm); Device: Sham Laser Therapy
- 650 nm LLLT (Salus Talent) (Experimental): Participants will receive low-level laser therapy using the Salus Talent device at a wavelength of 650 nm after complex decongestive physiotherapy (CDPT), which includes manual lymphatic drainage, remedial exercises, and intermittent pneumatic compression.
  Interventions: Device: Low-Level Laser Therapy (904 nm); Device: Sham Laser Therapy
- Sham Laser Therapy (Placebo Comparator): Participants will receive sham laser therapy with no active laser emission after complex decongestive physiotherapy (CDPT), which includes manual lymphatic drainage, remedial exercises, and intermittent pneumatic compression.
  Interventions: Device: Low-Level Laser Therapy (904 nm); Device: Low-Level Laser Therapy (650 nm)

INTERVENTIONS:
Device: Low-Level Laser Therapy (904 nm) — Low-level laser therapy using the LTU-904 device (RianCorp, Australia) at a wavelength of 904 nm, applied to the fibrotic area of the upper limb after CDPT.
  Arms: 650 nm LLLT (Salus Talent); Sham Laser Therapy
Device: Low-Level Laser Therapy (650 nm) — Low-level laser therapy using the Salus Talent device (Remed, USA) at a wavelength of 650 nm, applied to the fibrotic area of the upper limb after CDPT.
  Arms: 904nm LLLT (LTU-904); Sham Laser Therapy
Device: Sham Laser Therapy — Placebo laser therapy with no active laser emission, administered after CDPT.
  Arms: 650 nm LLLT (Salus Talent); 904nm LLLT (LTU-904)

SUMMARY:
This study is a prospective, single-blinded, randomized controlled trial designed to evaluate the effectiveness of low-level laser therapy (LLLT) using two different wavelengths (904 nm and 650 nm) in patients with secondary lymphedema following breast cancer surgery. Participants will be randomly assigned to one of three groups: 904 nm LLLT, 650 nm LLLT, or sham treatment. The primary objective is to assess changes in arm volume and secondary lymphedema-related outcomes following a structured intervention program.

DETAILED DESCRIPTION:
This single-blinded, parallel-group, randomized controlled trial will be conducted at a tertiary hospital. Eligible participants are women diagnosed with secondary lymphedema after breast cancer surgery. Patients with primary lymphedema, history of upper limb trauma, bilateral arm infection, or metastasis will be excluded. Participants will be randomized into three groups: Group A (904 nm LLLT), Group B (650 nm LLLT), and a sham group.

Each participant will receive ten treatment sessions. Every session will consist of 60 minutes of conventional complex decongestive physiotherapy (CDPT), including manual lymphatic drainage, remedial exercises, and intermittent pneumatic compression, followed by 20 minutes of laser therapy. All participants will receive fluoroscopy-guided manual lymphatic drainage during each session.

The 904 nm wavelength laser (LTU-904, RianCorp) and the 650 nm laser (Salus Talent, Remed) will deliver the same energy dose (22.5 J/cm²) during treatment. The sham group will receive placebo treatment with no active laser emission. Laser therapy will be applied to the most fibrotic area of the affected upper limb in a circular area approximately 7 cm in diameter. The irradiation will be performed point-by-point with 1 cm intervals. Five-minute rest intervals will be given between treatments.

Randomization will be conducted using stratified block randomization (block size of 4), and allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes. Participants will be blinded to the wavelength used. Outcome assessors will also be blinded to group allocation.

The primary outcome is change in upper limb volume. Secondary outcomes include changes in extracellular fluid ratio, tissue dielectric constant, circumferential measurements. Pre- and post-intervention assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Secondary lymphedema following breast cancer surgery

Exclusion Criteria:

* Primary lymphedema
* History of trauma, metastasis, or infection in both arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in subcutaneous tissue thickness of the affected upper limb | Baseline and after 10 sessions (approximately 3 weeks)
  Subcutaneous tissue thickness will be measured using B-mode ultrasonography (7.5 MHz linear-array transducer, Siemens Medical Solutions). Measurements will be taken at five predefined anatomical sites of the affected upper limb: (1) midpoint of the wrist crease, (2) medial epicondyle, (3) lateral epicondyle, (4) 10 cm proximal and distal to the elbow joint along predefined lines on both medial and lateral sides, and (5) the web space between the first and second fingers. Thickness values will be used to assess local soft tissue changes in response to treatment.
Change in dermal backflow (DB) pattern on indocyanine green (ICG) lymphography | Baseline and after 10 sessions (approximately 3 weeks)
  Indocyanine green (Diagnogreen, 2.5 mg/mL) will be injected intradermally into the first and third web spaces of the affected hand (0.1 mL per site). To minimize discomfort, lidocaine HCl 2% with epinephrine (1:100,000) will be administered prior to injection. Lymphatic flow will be visualized using near-infrared fluorescence imaging. Dermal backflow patterns will be classified from Type I to Type V according to established staging criteria, reflecting the severity and distribution of lymphatic stasis. The DB stage will be used as an indicator of lymphatic dysfunction and treatment response.

SECONDARY OUTCOMES:
Change in extracellular fluid (ECF) ratio | Baseline and after 10 sessions (approximately 3 weeks)
  ECF ratio will be assessed using multi-frequency bioimpedance analysis (MFBIA).
Change in upper limb volume | Baseline and after 10 sessions (approximately 3 weeks)
  Arm volume will be measured using standardized circumferential measurements and calculated using the truncated cone formula.

CONTACTS AND LOCATIONS:
Overall Officials: Jin A Yoon, MD, Ph.D, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, Seo-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed Omar MT, Abd-El-Gayed Ebid A, El Morsy AM. Treatment of post-mastectomy lymphedema with laser therapy: double blind placebo control randomized study. J Surg Res. 2011 Jan;165(1):82-90. doi: 10.1016/j.jss.2010.03.050. Epub 2010 Apr 18. PMID 20538293
- [Background] Jang DH, Song DH, Chang EJ, Jeon JY. Anti-inflammatory and lymphangiogenetic effects of low-level laser therapy on lymphedema in an experimental mouse tail model. Lasers Med Sci. 2016 Feb;31(2):289-96. doi: 10.1007/s10103-015-1854-y. Epub 2015 Dec 29. PMID 26714983
- [Background] Dirican A, Andacoglu O, Johnson R, McGuire K, Mager L, Soran A. The short-term effects of low-level laser therapy in the management of breast-cancer-related lymphedema. Support Care Cancer. 2011 May;19(5):685-90. doi: 10.1007/s00520-010-0888-8. Epub 2010 May 6. PMID 20445997
- [Background] Mayrovitz HN, Davey S. Changes in tissue water and indentation resistance of lymphedematous limbs accompanying low level laser therapy (LLLT) of fibrotic skin. Lymphology. 2011 Dec;44(4):168-77. PMID 22458118
- [Background] Berger AM, Mooney K, Alvarez-Perez A, Breitbart WS, Carpenter KM, Cella D, Cleeland C, Dotan E, Eisenberger MA, Escalante CP, Jacobsen PB, Jankowski C, LeBlanc T, Ligibel JA, Loggers ET, Mandrell B, Murphy BA, Palesh O, Pirl WF, Plaxe SC, Riba MB, Rugo HS, Salvador C, Wagner LI, Wagner-Johnston ND, Zachariah FJ, Bergman MA, Smith C; National comprehensive cancer network. Cancer-Related Fatigue, Version 2.2015. J Natl Compr Canc Netw. 2015 Aug;13(8):1012-39. doi: 10.6004/jnccn.2015.0122. PMID 26285247
- [Background] Buso G, Depairon M, Tomson D, Raffoul W, Vettor R, Mazzolai L. Lipedema: A Call to Action! Obesity (Silver Spring). 2019 Oct;27(10):1567-1576. doi: 10.1002/oby.22597. PMID 31544340
- [Background] Gustavsson S, Kelly KA, Hench VS, Melton LJ 3rd. Giant gastric and duodenal ulcers: a population-based study with a comparison to nongiant ulcers. World J Surg. 1987 Jun;11(3):333-8. doi: 10.1007/BF01658111. No abstract available. PMID 3604241
- [Background] Assis L, Moretti AI, Abrahao TB, de Souza HP, Hamblin MR, Parizotto NA. Low-level laser therapy (808 nm) contributes to muscle regeneration and prevents fibrosis in rat tibialis anterior muscle after cryolesion. Lasers Med Sci. 2013 May;28(3):947-55. doi: 10.1007/s10103-012-1183-3. Epub 2012 Aug 17. PMID 22898787
- [Background] Smoot B, Chiavola-Larson L, Lee J, Manibusan H, Allen DD. Effect of low-level laser therapy on pain and swelling in women with breast cancer-related lymphedema: a systematic review and meta-analysis. J Cancer Surviv. 2015 Jun;9(2):287-304. doi: 10.1007/s11764-014-0411-1. Epub 2014 Nov 29. PMID 25432632
- [Background] De Vrieze T, Vos L, Gebruers N, Tjalma WAA, Thomis S, Neven P, Nevelsteen I, De Groef A, Vandermeeren L, Belgrado JP, Devoogdt N. Protocol of a randomised controlled trial regarding the effectiveness of fluoroscopy-guided manual lymph drainage for the treatment of breast cancer-related lymphoedema (EFforT-BCRL trial). Eur J Obstet Gynecol Reprod Biol. 2018 Feb;221:177-188. doi: 10.1016/j.ejogrb.2017.12.023. Epub 2017 Dec 16. PMID 29277358
- [Background] Kilmartin L, Denham T, Fu MR, Yu G, Kuo TT, Axelrod D, Guth AA. Complementary low-level laser therapy for breast cancer-related lymphedema: a pilot, double-blind, randomized, placebo-controlled study. Lasers Med Sci. 2020 Feb;35(1):95-105. doi: 10.1007/s10103-019-02798-1. Epub 2019 May 11. PMID 31079232
- [Background] Szuba A, Shin WS, Strauss HW, Rockson S. The third circulation: radionuclide lymphoscintigraphy in the evaluation of lymphedema. J Nucl Med. 2003 Jan;44(1):43-57. PMID 12515876
- [Background] Unno N, Nishiyama M, Suzuki M, Tanaka H, Yamamoto N, Sagara D, Mano Y, Konno H. A novel method of measuring human lymphatic pumping using indocyanine green fluorescence lymphography. J Vasc Surg. 2010 Oct;52(4):946-52. doi: 10.1016/j.jvs.2010.04.067. PMID 20619581
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123
- [Background] Narushima M, Yamamoto T, Ogata F, Yoshimatsu H, Mihara M, Koshima I. Indocyanine Green Lymphography Findings in Limb Lymphedema. J Reconstr Microsurg. 2016 Jan;32(1):72-9. doi: 10.1055/s-0035-1564608. Epub 2015 Sep 30. PMID 26422172
- [Background] Yoon JA, Shin MJ, Shin YB, Kim K, Park H, Kang T, Kong IJ, Kim H, Park MS, Kim JH. Correlation of ICG lymphography and lymphoscintigraphy severity stage in secondary upper limb lymphedema. J Plast Reconstr Aesthet Surg. 2020 Nov;73(11):1982-1988. doi: 10.1016/j.bjps.2020.08.055. Epub 2020 Aug 25. PMID 32952056
- [Background] Niimi K, Hirai M, Iwata H, Miyazaki K. Ultrasonographic findings and the clinical results of treatment for lymphedema. Ann Vasc Dis. 2014;7(4):369-75. doi: 10.3400/avd.oa.14-00104. Epub 2014 Dec 25. PMID 25593621
- [Background] Lim CY, Seo HG, Kim K, Chung SG, Seo KS. Measurement of lymphedema using ultrasonography with the compression method. Lymphology. 2011 Jun;44(2):72-81. PMID 21949976
- [Background] Polat AV, Ozturk M, Polat AK, Karabacak U, Bekci T, Murat N. Efficacy of Ultrasound and Shear Wave Elastography for the Diagnosis of Breast Cancer-Related Lymphedema. J Ultrasound Med. 2020 Apr;39(4):795-803. doi: 10.1002/jum.15162. Epub 2019 Nov 9. PMID 31705687
- [Background] Cornish BH, Thomas BJ, Ward LC. Improved prediction of extracellular and total body water using impedance loci generated by multiple frequency bioelectrical impedance analysis. Phys Med Biol. 1993 Mar;38(3):337-46. doi: 10.1088/0031-9155/38/3/001. PMID 8451277
- [Background] Bae SH, Kim WJ, Seo YJ, Kim J, Jeon JY. Bioimpedance Analysis for Predicting Outcomes of Complex Decongestive Therapy for Gynecological Cancer Related Lymphedema: A Feasibility Study. Ann Rehabil Med. 2020 Jun;44(3):238-245. doi: 10.5535/arm.19102. Epub 2020 Jun 30. PMID 32640783
- [Background] Mayrovitz HN. Assessing local tissue edema in postmastectomy lymphedema. Lymphology. 2007 Jun;40(2):87-94. PMID 17853619
- [Background] Barbosa RI, Guirro ECO, Bachmann L, Brandino HE, Guirro RRJ. Analysis of low-level laser transmission at wavelengths 660, 830 and 904 nm in biological tissue samples. J Photochem Photobiol B. 2020 Aug;209:111914. doi: 10.1016/j.jphotobiol.2020.111914. Epub 2020 May 22. PMID 32516626
- [Background] Carati CJ, Anderson SN, Gannon BJ, Piller NB. Treatment of postmastectomy lymphedema with low-level laser therapy: a double blind, placebo-controlled trial. Cancer. 2003 Sep 15;98(6):1114-22. doi: 10.1002/cncr.11641. PMID 12973834
- [Background] Wang Y, Ge Y, Xing W, Liu J, Wu J, Lin H, Lu Y. The effectiveness and safety of low-level laser therapy on breast cancer-related lymphedema: An overview and update of systematic reviews. Lasers Med Sci. 2022 Apr;37(3):1389-1413. doi: 10.1007/s10103-021-03446-3. Epub 2021 Nov 15. PMID 34779937
- [Background] E Lima MT, E Lima JG, de Andrade MF, Bergmann A. Low-level laser therapy in secondary lymphedema after breast cancer: systematic review. Lasers Med Sci. 2014 May;29(3):1289-95. doi: 10.1007/s10103-012-1240-y. Epub 2012 Nov 29. PMID 23192573
- [Background] Baxter GD, Liu L, Petrich S, Gisselman AS, Chapple C, Anders JJ, Tumilty S. Low level laser therapy (Photobiomodulation therapy) for breast cancer-related lymphedema: a systematic review. BMC Cancer. 2017 Dec 7;17(1):833. doi: 10.1186/s12885-017-3852-x. PMID 29216916
- [Background] Lahtinen T, Seppala J, Viren T, Johansson K. Experimental and Analytical Comparisons of Tissue Dielectric Constant (TDC) and Bioimpedance Spectroscopy (BIS) in Assessment of Early Arm Lymphedema in Breast Cancer Patients after Axillary Surgery and Radiotherapy. Lymphat Res Biol. 2015 Sep;13(3):176-85. doi: 10.1089/lrb.2015.0019. Epub 2015 Aug 25. PMID 26305554